CLINICAL TRIAL: NCT01879956
Title: Randomized Controlled Trial for the Evaluation of the Efficacy of Occupational Therapy in the Rehabilitation of Executive Functions in Patients With Refractory Schizophrenia
Brief Title: Occupational Therapy in the Rehabilitation of Executive Functions in Patients With Schizophrenia
Acronym: OTSchizo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Helio Elkis, Associate Professor of the Department of Psychiatry, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OT Schizophrenia_1
Record Dates: First submitted 2013-05-29; First posted 2013-06-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Refractory Schizophrenia
Keywords: Executive Functions; Schizophrenia; Occupational Therapy
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant; Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OGI Method (Active Comparator): - experimental group: use the OGI method to improve the executive functioning of patients with refractory schizophrenia.
  Interventions: Behavioral: OGI Method
- craft activities (Placebo Comparator): - control group: use of craft activities, attend the same-number of sessions, but without the intervention of therapists.
  Interventions: Other: Craft Activities

INTERVENTIONS:
Other: Craft Activities — There is no intervention method used to perform the task.
  Arms: craft activities
Behavioral: OGI Method — metacognitive approach to assess executive functions.
  Arms: OGI Method

SUMMARY:
Primary Objective:

Efficacy of Occupational Therapy (OT) based Occupational Goal Intervention (OGI) in improving executive functions in patients with refractory schizophrenia as measured by the BADS.

Secondary Objectives: improvement of functional aspects,basic and instrumental activities of daily living,negative symptoms and cognitive functions improvement

Hypothesis: OT is more effective than control group to improve executive functions in patients with refractory schizophrenia.

DETAILED DESCRIPTION:
A single-center, randomized, single blind, controlled study, lasting one year, including the follow-up.

The study is conducted in two groups:the experimental group is based on the OGI method (N=30 patients) and the control group receives craft activities (N = 30 patients).

Psychiatric, neuropsychological and functional aspects are assessed at the beginning, after 30 sessions and 6 months after the intervention. The scale PANSS (Positive and Negative Syndrome Scale) is used for monitoring psychopathological symptoms during the study.

Scales BADS, DAFS-R, ILSS-BR respectively assess executive functions, functionality and basic and instrumental activities of daily living. The neuropsychological evaluation includes a battery to measure attention, executive functions, memory and estimated intellectual efficiency.

Statistical analysis to be used: ANOVA (Analysis of Variance)for repeated measures; data are also calculated to messure clinical efficacy, effect size and needed number to treat.

ELIGIBILITY:
Inclusion Criteria:

* Pacients with diagnosis of schizophrenia for DMS IV-R.
* Pacients that signed the consent in writing and receive explanations about the nature of the study.
* Patients who carefully counted another responsible person to provide reliable support to the patient and ensure adherence to the same study treatment.
* Patients with minimum education: five years (elementary school).

  * Patients who present rates below those expected for their age group in at least 3 of the executive functions assessed on neuropsychological tests, and evaluation of executive functions.
* Patients with stable clozapine and which have not been recently admitted (3 months).

Exclusion Criteria:

* Comorbid diagnosis of substance dependence or other psychiatric Axis I;
* History of head trauma and / or other neurological problems;
* Medical problems that compromise somehow the central nervous system;
* History of mental retardation;
* Patients treated with medication other than clozapine;
* Patients who are suffering other psychosocial treatments.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
BADS (Behavioral Assessment of Functional Status) | up to 6 months follow-up.
  It is a battery which measures neuropsychological executive functions.

SECONDARY OUTCOMES:
DAFS-BR ( Direct Assessment of Functional Status), ILSS-BR (Habilities of Daily Living-Brazilian validated version). | at baseline, after 30 sessions of treatment and follow-up 6 months.
  DAFS-BR - Evaluates functional aspects of daily living such as dealing with money, shopping, social comunication ILSS-BR- similar to DAFS.
Trail Making A/B, Digit Span, Wisconsin Card Sorting Test, Stroop Color Test, Rey Complex Figure, Verbal Fluency,Tapping Visual and Logical Memory. | at baseline, after 30 sessions of treatment and 6 months follo-up.
  Neuropsychological Battery (Trail Making A/B, Digit Span, Wisconsin Card Sorting Test, Stroop Color Test,Rey Complex Figure, Fluência Verbal, Tapping Visual and Memória Logica)which measure cognitive functions.
Trail Making A/B, Digit Span, Wisconsin Card Sorting Test, Stroop Color Test, Rey Complex Figure, Verbal Fluency,Tapping Visual and Logical Memory. | at baseline, after 30 sessions of treatment and 6 months follo-up.
  Neuropsychological Battery (Trail Making A/B, Digit Span, Wisconsin Card Sorting Test, Stroop Color Test,Rey Complex Figure, Verbal Fluency, Tapping Visual and Memória Logica)which measure cognitive functions.

CONTACTS AND LOCATIONS:
Overall Officials: Helio Elkis, MD PhD, Principal Investigator — Departamento de Psiquiatria da FMUSP
Locations (1):
- Instituto de Psiquiatria do HCFMUSP, São Paulo, São Paulo, Brazil